CLINICAL TRIAL: NCT01597219
Title: A UK Multicentre Study of Haploidentical Stem Cell Transplantation in Patients With Haematological Malignancies
Brief Title: Trial of Haploidentical Stem Cell Transplantation for Haematological Cancers
Acronym: UK-Haplo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Bloodwise (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/10/0411
Record Dates: First submitted 2012-05-10; First posted 2012-05-11 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Acute Myeloid Leukaemia; Acute Lymphoblastic Leukaemia; Myelodysplastic Syndrome; Chronic Myeloid Leukaemia; Chronic Lymphocytic Leukaemia; Acquired Bone Marrow Failure Syndromes; Other Haematological Malignancies; Unrelated HSCT Indicated
Keywords: Haploidentical transplant; Haematological malignancy; Myeloablative; Reduced intensity
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, B-Cell; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced intensity haploidentical transplant (Experimental): Fludarabine 30mg/m2 IV days -6 to -2 Cyclophosphamide 14.5 mg/kg IV days -6 and -5 Total body irradiation 2Gy day -1 Stem cell transplant: day 0 Cyclophosphamide 50mg/kg days +3 & +4
  Interventions: Procedure: Reduced intensity haplodentical stem cell transplant
- Myeloablative haploidentical stem cell transplant (Experimental): Total body irradiation 12Gy in 8 fractions days -9 to -6 Donor lymphocyte infusion day -6 Cyclophosphamide 60mg/kg IV days -3 & -2 Stem cell transplant day 0
  Interventions: Procedure: Myeloablative haploidentical stem cell transplant

INTERVENTIONS:
Procedure: Reduced intensity haplodentical stem cell transplant — Fludarabine 30mg/m2 IV days -6 to -2 Cyclophosphamide 14.5 mg/kg IV days -6 and -5 Total body irradiation 2Gy day -1 Stem cell transplant: day 0 Cyclophosphamide 50mg/kg days +3 & +4
  Arms: Reduced intensity haploidentical transplant
Procedure: Myeloablative haploidentical stem cell transplant — Total body irradiation 12Gy in 8 fractions days -9 to -6 Donor lymphocyte infusion day -6 Cyclophosphamide 60mg/kg IV days -3 & -2 Stem cell transplant day 0
  Arms: Myeloablative haploidentical stem cell transplant

SUMMARY:
This trial investigates stem cell transplants from partially mismatched donors in patients with blood and bone marrow cancers. The trial will test two kinds of transplants - a full intensity transplant using a high dose of radiotherapy and chemotherapy, and a reduced intensity transplant with lower doses of chemotherapy and radiotherapy. Patients will be entered for the treatment pathway that is most appropriate for their level of health and fitness

ELIGIBILITY:
Patient Inclusion Criteria

1. Eligible for an allogeneic transplant in line with the current BSBMT indications for transplant criteria (http://bsbmt.org/indications-table/) accepted by Commissioners
2. Age 16-70
3. Adequate physical function

   * Cardiac: LVEF at rest ≥45%, or shortening fraction ≥25%
   * Hepatic: Bilirubin ≤35mmol/l; AST/ALT and alkaline phosphatase <5 x ULN
   * Renal: Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, creatinine clearance or GFR >40ml/min/1.73m2
   * Pulmonary: FEV1, FVC, DLCO (diffusion capacity) >50% predicted (corrected for haemoglobin); if clinically unable to perform pulmonary function tests then O2 saturation >92% on room air
   * Performance status: Karnofsky score ≥60%
4. Donor available aged ≥16 years
5. Needs an urgent transplant where a 10/10 HLA matched sibling or unrelated donor is unavailable in a timely manner. An unrelated donor search is not required for a patient to be eligible if the clinical situation dictates an urgent transplant. Clinical urgency is defined as 6-8 weeks from referral to transplant centre or low likelihood of finding a matched unrelated donor
6. HLA typing will be performed at high resolution (allelic) for the HLA-A, HLA-B, HLA-Cw, HLA-DRB1 and HLA-DQB1 loci. A minimum match of 5/10 is required
7. The donor and recipient must be identical as determined by high resolution typing at at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1 and HLA-DQB1. Fulfilment of this criterion is sufficient evidence that the donor and recipient share one HLA haplotype and typing of additional family members is not required.
8. Patient must have received cytotoxic chemotherapy within 3 months of the consent date (measured from the start date of the most recent cycle of chemotherapy) except patients with aplastic anaemia, unless otherwise agreed by the TMG (see section 5.3.4). The use of monoclonal antibody therapy may be considered cytotoxic chemotherapy, but must be agreed by the TMG
9. Written informed consent

Donor Inclusion Criteria

1. Donor must be an HLA-haploidentical first degree relative of the patient. Eligible donors include biological parents, siblings, children or half-siblings
2. Age ≥16 years
3. Donors must meet the collection centre's usual selection criteria for related allogeneic HPC donors

Patient Exclusion Criteria

1. HLA matched, related donor able to donate
2. Autologous haematopoietic stem cell transplant <3 months prior to enrolment
3. Pregnancy or breastfeeding
4. Uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiological findings), the inclusion of patients with an uncontrolled viral or fungal infection can be agreed by the TMG
5. Serious psychiatric or psychological disorders
6. Absence or inability to provide informed consent
7. Severe comorbidity (HCT-CI comorbidity score of 3 or more) or disease that prevents treatment with chemotherapy, unless otherwise agreed by the TMG
8. Positive anti-donor HLA antibody
9. Unable to receive 2Gy TBI (RIC pathway) or 12Gy TBI (MAC pathway)
10. Patients with graft rejection following a previous allograft from either adult or cord blood donors

Donor Exclusion Criteria

1. Positive anti-donor HLA antibody in the recipient
2. Pregnancy or recent birth (within 6 months prior to donating cells)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-03; Primary Completion 2024-01 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kavita Raj, Principal Investigator — King's College Hospital NHS Trust
Locations (12):
- United Kingdom (12):
  - Birmingham Heartlands, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Beatson Hospital, Glasgow
  - St James' University Hospital, Leeds
  - Royal Liverpool Hospital, Liverpool
  - King's College Hospital, London
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle
  - Royal Hallamshire, Sheffield & Weston Park, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided